CLINICAL TRIAL: NCT06954844
Title: tVNS to Provide Mechanistic Insights Into the Relationship Between Systemic Inflammation and Altered Motivation and Mood in Healthy Individuals Who Are Overweight or Obese
Brief Title: tVNS and Obesity-related Mechanisms
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bonn (Other)
Responsible Party: Principal Investigator, Dr. Nils B. Kroemer, Prof. Dr. rer. nat., University Hospital, Bonn
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: BON006; 493623632 (Other Grant/Funding Number: Deutsche Forschungsgemeinschaft (DFG, German Research Foundation))
Record Dates: First submitted 2025-03-21; First posted 2025-05-02 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Overweight/Obesity (BMI: 27 and 35 kg/m2)
Keywords: Inflammation; Metaflammation; tVNS; Motivation
MeSH Terms: conditions — Overweight; Obesity; Inflammation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity transcutaneous non-invasive vagus nerve stimulation (tVNS) (Experimental): Participants will receive high intensity tVNS for >30 min per day for 14 days at home. To stimulate vagal afferents, the electrode will be placed at the cymba conchae of the right ear using a previously established conventional stimulation protocol (30 s ON, 30s OFF, 25 Hz frequency, 250 µs pulse widths; tVNS R device, tVNS Technologies GmbH, Erlangen, Germany). Stimulation intensity will be pre-set for each participant for the following stimulation period to correspond to a mild pricking sensation determined with a staircase procedure in the lab session.
  Interventions: Device: Transcutaneous non-invasive vagus nerve stimulation (tVNS)
- Low intensity stimulation (Sham Comparator): The control intervention consists of low intensity stimulation. Participants will receive low intensity stimulation for >30 min per day for 14 days at home. The electrode will be placed at the cymba conchae, but only receive a low-intensity stimulation below the perception threshold (0.1mA, 1s ON, 30s OFF, 1 Hz frequency, 250 µs pulse widths; tVNS R device, tVNS Technologies GmbH, Erlangen, Germany).
  Interventions: Device: Low intensity stimulation

INTERVENTIONS:
Device: Transcutaneous non-invasive vagus nerve stimulation (tVNS) — To stimulate vagal afferents, the electrode will be placed at the cymba conchae of the right ear using a previously established conventional stimulation protocol (30 s ON, 30s OFF, 25 Hz frequency, 250 µs pulse widths; tVNS R device, tVNS Technologies GmbH, Erlangen, Germany). Stimulation intensity will be pre-set for each participant for the following stimulation period to correspond to a mild pricking sensation determined with a staircase procedure in the lab session.
  Arms: High intensity transcutaneous non-invasive vagus nerve stimulation (tVNS)
Device: Low intensity stimulation — The electrode will be placed at the cymba conchae, but only receive a low-intensity stimulation below the perception threshold (0.1mA, 1s ON, 30s OFF, 1 Hz frequency, 250 µs pulse widths; tVNS R device, tVNS Technologies GmbH, Erlangen, Germany).
  Arms: Low intensity stimulation

SUMMARY:
The overarching goal of the project is to assess whether transcutaneous Vagus Nerve Stimulation (tVNS) induced reduction of central and peripheral inflammation is associated with tVNS induced changes in mood and motivation in a sample of healthy participants with overweight and obesity.

DETAILED DESCRIPTION:
Participants will receive high intensity or low intensity tVNS in a single-blind, randomized, crossover design. Each stimulation (high and low intensity) will be applied over 14 days (effective minimum duration) at home by the participants, with a 7-day (effective minimum duration) washout period in between the conditions. To assess the effect of high (vs. low intensity) stimulation on inflammation and mood/motivation, the investigators plan to use a combination of blood analysis, ecological momentary assessments (EMA), and neuroimaging sessions. To this end, the investigators will apply functional Magnetic Resonance Imaging (fMRI), diffusion basis spectrum imaging (DBSI), and a behavioural task capturing different facets of motivation. During the study, participants will be invited for four lab-based sessions (t0-t3). The first visit before the start of the stimulation (t0) will be used to measure baseline levels of mood, motivation, and inflammation, as well as body measures, and metabolic blood parameter. Additionally, participants will be asked to rate standardized food pictures for liking, wanting, healthiness, and environmental sustainability during the first lab-based session (t0). These ratings will be used for a food choice task during the intervention phase, which is described in more detail below. To track changes induced by the intervention, the second (t1) and fourth visits (t3) will take place after 14 days of daily stimulation with high or low intensity stimulation, respectively. There will be a 7-day washout period in between the end of the first stimulation phase and the start of the second. In the third session (t2), participants will be instructed how to use the tVNS device in the crossover condition at home and mood, body measures, and metabolic blood parameter will be measured again before the second intervention phase. The third session will take place after the 7-day washout period.

Sessions at t0, t1, and t3: Participants will be asked to come in a fasted (12h) state. After a short mood and metabolic state survey (Positive and Negative Affect Schedule (PANAS) items presented on a visual analogue scale (VAS) on a computer), the investigators will determine resting heart rate, blood pressure, and body measures (such as body height, weight and percentage of body fat). A blood sample will then be taken to measure peripheral inflammation (cytokines, circulating blood cells) and metabolic parameter (insulin sensitivity, blood lipid levels). Subsequently, the participants will perform an effort allocation task (EAT) during fMRI. In the EAT, participants are asked to move a ball above a drawn line (representing the difficulty) by exerting effort (e.g., by rapidly pressing a button or a grip force handle inside the scanner) to collect different types of reward (food and money). Trials within the task vary in difficulty, reward type (food vs. money), and reward magnitude (1 point vs. 10 points). After each trial, participants are asked to rate how much they wanted the reward and how much they exerted effort during the trial. In addition, a diffusion-weighted sequence is acquired in the MRI to measure central inflammation. The investigators will then assess mood (PANAS items) again and participants will be instructed to use the device for >30 min per day at home (stimulation use will be logged by the devices). After the session participants will be paid out the rewards gained during the task. 80% of the calories are paid out as breakfast (muesli with milk) and 20% of the calories as snacks (e.g. chocolate, wine gums). After paying out the rewards gained during the task, the investigators will again assess mood, using the PANAS items.

Sessions at t2: Participants will be asked to come in a fasted (12h) state. After a short mood and metabolic state survey (PANAS items presented on a visual analogue scale (VAS) on a computer), the investigators will determine resting heart rate, blood pressure, and body measures. A blood sample will then be taken to measure metabolic parameter (insulin sensitivity, blood lipid levels). Participants will then be instructed how to use the tVNS device in the crossover condition at home. Afterwards, the investigators will again assess mood, using the PANAS items.

During the intervention phases, Ecological momentary assessments (EMA) (e.g., "how happy do you feel at the moment?", "how sad do you feel at the moment?", and "how motivated do you feel right now?") will be completed daily. In addition, EMA questions will be used to assess subjective control over eating behaviour (e.g., "While you were eating, to what extent did you feel a sense of loss of control?" and physical activity ("How many minutes of moderate or strenuous physical activity did you do today?"). A food choice task will be used to assess changes in eating behaviour. Therefore, participants will be asked to rate standardized food pictures for liking, wanting, healthiness, and environmental sustainability during the first lab-based session (t0). A choice task will be used to assess changes in decision weights. Two pictures that have been rated similarly for one domain (e.g. liking) will be presented to the participants, who will be instructed to choose one of the pictures. Decisions will be used to estimate decision weights for the remaining three domains.

Standardized questionnaires will be used to characterize our sample. The investigators will e.g., assess symptoms of depression, anhedonia, and apathy (Becks Depression Inventory, (BDI-II), Snaith-Hamilton Please Scale in German (SHAPS-D), and Apathy Motivation Index (AMI)). Additionally, the investigators will assess eating behaviour (using a food frequency questionnaire from the "German Health Interview and Examination Survey for Adults 2008-2011" (DEGS)), as well as physical activity (International Physical Activity Questionnaire (IPAQ)).

Five major hypotheses will be tested:

Hypothesis 1: Participants will have lower levels of peripheral inflammation measured as reduced levels of pro-inflammatory cytokines, enhanced levels of anti-inflammatory cytokines, and changes in the circulating immune cells after high compared to low intensity stimulation.

Hypothesis 2: Participants will have reduced central inflammation reflected in reduced tissue edema and cellularity after high compared to low intensity stimulation.

Hypothesis 3: Participants will have improved mood (as measured by items of the Positive and Negative Affect Schedule; PANAS) after high compared to low intensity stimulation.

Hypothesis 4: Participants will have enhanced motivation to work for rewards after high compared to low intensity stimulation.

Hypothesis 5: The tVNS-induced (high vs. low intensity) reduction of central and peripheral inflammation is associated with tVNS-induced changes in mood and motivation.

Secondary hypotheses:

Hypothesis 6: Levels of peripheral and central inflammation are associated with mood and motivation

Hypothesis 7: Participants will have enhanced ratings of reward wanting during the EAT after high compared to low intensity stimulation.

Hypothesis 8: Participants will have decreased utility slopes in the EAT after high compared to low intensity stimulation.

Hypothesis 9: Participants will have improved mood and motivation measured using EMA questions during high intensity stimulation phases compared to low intensity stimulation phases.

Hypothesis 10: Participants will show reduced anhedonia after high compared to low intensity stimulation.

Hypothesis 11: Participants will show reduced depressive symptoms after high compared to low intensity stimulation.

Hypothesis 12: Participants will show reduced apathy after high compared to low intensity stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 40 years of age
* BMI between 27 and 35.0 kg/m2
* Legally valid declaration of consent

Exclusion Criteria:

* Current or past diagnosis of brain injury/surgery or neurological condition with permanent effects, epilepsy, stroke, schizophrenia, bipolar disorder, severe substance use disorder, heart disease that precludes use of tVNS, diabetes (type 1 or 2), chronic inflammatory diseases (e.g., rheumatoid arthritis, Crohn's disease, etc.)
* Following diagnosis within 12 months before start of experiment: obsessive compulsive disorder, somatic symptom disorder, eating disorder
* Considerable weight change (>10%) within the last 6 months before the experiment
* Elevated BMI is due to fat-free mass (e.g., in athletes)
* Medication or Electroconvulsive therapy to treat a mental, metabolic, or neurological disorder (e.g., selective serotonin reuptake inhibitors, Glucagon-like Peptide-1 agonists) currently or in the last 3 months (hormone treatments that normalize function are not excluded)
* Anti-inflammatory medication currently or in the last 3 month
* Contraindications for MRI (e.g., metal implants, claustrophobia)
* Contraindications for tVNS (e.g., piercings, sore or diseased skin areas on the outer right ear)
* active implants (e.g., pacemaker), cerebral shunt
* Pregnant and breastfeeding women

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Stimulation-induced mid-term changes in a multiplex panel of different inflammatory biomarkers (peripheral inflammation) | Baseline, immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  To measure peripheral inflammation, the investigators will assess plasma levels of pro- and anti-inflammatory cytokines, chemokines, and other biomarker of inflammation (e.g. Growth Factors) using highly sensitive immunoassays (e.g. NULISA). The investigators will select the specific panel after data collection is complete and before data analysis begins, based on the literature and the analysis methods available at that time. Blood levels will be assessed at baseline and after each stimulation phase (high and low intensity; 14 days stimulation each). Multivariate analysis will be used to compare stimulation-induced changes in plasma levels between high and low intensity stimulation.
Stimulation-induced mid-term changes in circulating immune cells (peripheral inflammation) | Baseline, immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  To measure peripheral inflammation, the investigators will measure the following circulating immune cells using fluorescence flow cytometry: Leukocytes, lymphocytes, neutrophil granulocytes, T-cells, (Cluster of Differentiation (CD)4+, CD8+), naïve T cells (CD4+, CD8+), central memory T-cells (CD4+, CD8+), effector memory T-cells (CD4+, CD8+), terminal effector memory re-expressing CD45RA T cells, regulatory T cells (Treg) (activated, resting), conventional T cells, cytotoxic T-cells, T helper cells (Th), Th1 cells, Th2 cells, Th1/17 cells, Th17 cells, effector T-cells, mononuclear phagocytes, monocytes (classical, Intermediate, non-classical), dendritic cells (type 1 conventional, type 2 conventional, plasmacytoid). Cells will be assessed at baseline and after each stimulation phase (high and low intensity; 14 days stimulation each). Multivariate analysis will be used to compare stimulation-induced changes in circulating immune cells between high and low intensity stimulation.
Stimulation-induced mid-term changes in tissue edema as assessed using non-restricted fraction (isotropic DBSI-NRF (f(D), D = 0.3 - 3.0 μm2/ms)) | Baseline, immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  One measure of central inflammation will be the non-restricted fraction in the brain. This will be calculated with diffusion tensor imaging (DTI) measurement acquired with a 3 Tesla (3T) Siemens Scanner. Non-restricted fraction is calculated as the isotropic DBSI-NRF (f(D), D = 0.3 - 3.0 μm2/ms) and indicates tissue edema. Regions of interest (ROI) will be defined using the Harvard Oxford extended Atlas and include the putamen, caudate, pallidum, and nucleus accumbens (NAcc) as well as the hypothalamus. Non-restricted fraction will be assessed at baseline and after each stimulation phase (high and low intensity; 14 days stimulation each) and compared in predefined ROIs between high and low intensity stimulation.
Stimulation-induced mid-term changes in tissue cellularity as assessed using restricted fraction (isotropic DBSI-RF (f(D), D ≤ 0.3 μm2/ms)) | Baseline, immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  Another measure of central inflammation will be restricted fraction indicating tissue cellularity. This will be calculated with diffusion tensor imaging (DTI) measurement acquired with a 3T Siemens Scanner. Restricted fraction will be calculated as the isotropic DBSI-RF (f(D), D ≤ 0.3 μm2/ms) and indicates tissue edema. Regions of interest (ROI) will be defined using the Harvard Oxford extended Atlas and include the putamen, caudate, pallidum, and NAcc as well as the hypothalamus. Restricted fraction will be assessed at baseline and after each stimulation phase (high and low intensity; 14 days stimulation each) and compared in predefined ROIs between high and low intensity stimulation.
Stimulation-induced mid-term changes in PANAS items (mood) | Baseline (immediately before each stimulation phase), immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  To measure mood, the investigators will use items from the PANAS, rated on visual analogue scales (VAS) ranging from 0 (lowest rating) to 100 (highest rating). These items will be assessed at baseline (before each stimulation phase) and after each stimulation phase (high and low intensity; 14 days stimulation each). Values from the Positive and Negative Affect Schedule will be analysed as repeated measures assessing either positive (PA) or negative (NA) affect. Stimulation-induced changes in mood state (PA - NA) will be compared between high and low intensity stimulation.
Stimulation-induced mid-term changes in Invigoration (motivation) | Baseline, immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  Invigoration will be assessed using the effort allocation task and is captured by the slope of the initial approach (i.e., the increase of force until a first plateau is reached). Invigoration will be assessed at baseline and after each stimulation phase (high and low intensity; 14 days stimulation each). Stimulation-induced changes in Invigoration will be compared between high and low intensity stimulation.
Stimulation-induced mid-term changes in maintenance (motivation) | Baseline, immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  Maintenance will be assessed using the effort allocation task and reflects the average relative force/frequency across the whole trial. Maintenance will be assessed at baseline and after each stimulation phase (high and low intensity; 14 days stimulation each). Stimulation-induced changes in maintenance will be compared between high and low intensity stimulation.
Stimulation-induced mid-term changes in anticipatory neural reward response (motivation) | Baseline, immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  To evaluate anticipatory neural reward response, the investigators will assess fMRI bold signals during cue presentation prior to exerting effort during the effort allocation task using a 3T Siemens Scanner. The contrast of interest will be the modulation of the anticipatory response by the reward magnitude (high vs. low) combining responses to food and monetary rewards. Other contrasts (cue response itself and contrasts specific for food or monetary rewards are exploratory). Regions of Interest (ROI) will be defined using the Harvard Oxford extended Atlas. Primary ROIs will be the NAcc and ventromedial prefrontal cortex (vmPFC) and secondary ROIs will be ventral tegmental area (VTA)/substantia nigra (SN), and caudate, and putamen. fMRI metrics will be assessed at baseline and after each stimulation phase (high and low intensity; 14 days stimulation each). Stimulation-induced changes in bold signals in predefined ROI will be compared between high and low intensity stimulation.
Stimulation-induced mid-term changes in neural motor response (motivation) | Baseline, immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  To evaluate neural motor response, the investigators will assess fMRI bold signals while the participants exert effort (work phase) during the effort allocation task using a 3T Siemens Scanner. The contrasts of interest will be force/repetition time (TR) to assess motor work during the task and the first derivative of force/TR (temporal relative = d(force)/d(TR)) estimating the drive to work. Region of Interest (ROI) will be defined using the Harvard Oxford extended Atlas and include the supplementary motor area (SMA) and pre-SMA, as well as VTA/SN, and caudate, putamen, and NAcc. fMRI metrics will be assessed at baseline and after each stimulation phase (high and low intensity; 14 days stimulation each). Stimulation-induced changes in bold signals in predefined ROI will be compared between high and low intensity stimulation.
Correlation of Stimulation-induced changes in peripheral and central inflammation with changes in mood and motivation | Baseline, immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  The investigators will correlate changes (i.e., random effect estimates of high intensity stimulation slopes relative to low intensity stimulation) in peripheral and central inflammation markers with tVNS-induced (high vs. low intensity) changes in mood and motivation.

SECONDARY OUTCOMES:
Stimulation-induced mid-term changes in ratings of reward wanting and exertion | Baseline, immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  Ratings of wanting and exertion after each trial (after the effort exertion phase) in the effort allocation task will be assessed on a visual analogue scale ranging from 0 (lowest rating) to 100 (highest rating). Stimulation-induced changes in ratings will be compared between high and low intensity stimulation.
  Note: Exertion and wanting ratings are only assessed while participants perform the EAT outside the MRI, prior to the MRI task.
Stimulation-induced mid-term changes in utility slope | Baseline, immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  To investigate the correspondence between effort and wanting, the investigators will calculate "utility slopes" as the correlation between trial-wise wanting ratings and trial-wise effort maintenance. Stimulation-induced changes in utility slopes will be compared between high and low intensity stimulation.
  Note: Exertion and wanting ratings are only assessed while participants perform the EAT outside the MRI, prior to the MRI task.
Stimulation-induced changes in mood and motivation in daily life | During intervention phase: 14 days
  Mood and motivation will be assessed daily during the intervention phase via visual analogue scales ranging from 0 (lowest rating) to 100 (highest rating) using EMA. The main outcomes include mood assessed using mood state: (Happy - Sad)/100 and motivation (single item).
  List of items:
  How happy do you feel at the moment? How sad do you feel at the moment? How motivated do you feel right now?
  Stimulation-induced changes in mood and motivation ratings during the intervention phase will be compared between high and low intensity stimulation.
Stimulation-induced mid-term changes in anhedonia | Baseline, immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  The German version of the Snaith Hamilton Pleasure Scale (SHAPS-D) will be used to assess anhedonia at baseline and after each stimulation phase (high and low intensity; 14 days stimulation each). The questionnaire consists of four domains. The investigators will determine an overall outcome measure "anhedonia" using the sum score across all items (0-14), with higher scores indicating more severe anhedonia. This sum score will be used to compare changes induced by high vs low intensity stimulation.
Stimulation-induced mid-term changes in depressive symptoms | Baseline, immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  The Beck's Depression Inventory (BDI-II) will be used to assess changes in depressive symptoms at baseline and after each stimulation phase (high and low intensity; 14 days stimulation each). The items of the score will be summed up to a total score (0-63), with higher scores indicating more severe depression. This score will be used to compare changes induced by high vs. low intensity stimulation.
Stimulation-induced mid-term changes in apathy | Baseline, immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  The Apathy Motivation Index (AMI) will be used to assess apathy at baseline and after each stimulation phase (high and low intensity; 14 days stimulation each). The questionnaire consists of three subscales that can be combined to a total score (0-72), with higher scores indicating more severe apathy. The investigators will determine an overall outcome measure "apathy" using the sum score across all items to compare changes induced by high vs. low intensity stimulation.

OTHER OUTCOMES:
BMI | Baseline (immediately before each stimulation phase), immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  BMI (kg/m2) will be measured at baseline (before each stimulation phase) and after each stimulation phase (high and low intensity; 14 days stimulation each). Stimulation-induced changes will be compared between high and low intensity stimulation.
Percentage of body-fat | Baseline, immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  Percentage of body-fat will be measured at baseline and after each stimulation phase (high and low intensity; 14 days stimulation each). Stimulation-induced changes will be compared between high and low intensity stimulation.
Waist-to-hip ratio | Baseline (immediately before each stimulation phase), immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  Waist-to-hip ratio will be measured at baseline (before each stimulation phase) and after each stimulation phase (high and low intensity; 14 days stimulation each). Stimulation-induced changes will be compared between high and low intensity stimulation.
Eating behaviour | Baseline, immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  Eating behaviour will be evaluated using a food frequency questionnaire (FFQ) that was used in the "German Health Interview and Examination Survey for Adults 2008-2011" (DEGS) to evaluate the last 14 days. This food frequency questionnaire is used to enquire about the frequency of consumption and usual portion sizes of a total of 53 food groups consumed. Eating behaviour will be assessed at baseline and after each stimulation phase (high and low intensity; 14 days stimulation each). Stimulation-induced changes in questionnaire scores in food groups will be compared between high and low intensity stimulation using multivariate analysis.
Physical activity (1) | Baseline, immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  Participants will complete the long version of the International Physical Activity Questionnaire (IPAQ) to assess physical activity in the last 14 days at baseline and after each stimulation phase (high and low intensity; 14 days stimulation each). Stimulation-induced changes in questionnaire scores (e.g. metabolic equivalent (MET)-minutes/week) will be compared between high and low intensity stimulation.
Physical activity (2) | During intervention phase: 14 days
  EMA will be used to assess the number of minutes of moderate and strenuous physical activity daily during the intervention phase. Stimulation-induced changes in minutes of physical activity during the intervention phase will be compared between high and low intensity stimulation.
  Item:
  How many minutes of moderate or strenuous physical activity did you do today?
Stimulation-induced mid-term changes in fat metabolism | Baseline (immediately before each stimulation phase), immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  High Density Lipoprotein (HDL), Low Density Lipoprotein (LDL), and LDL/HDL quotient will be assessed at baseline (before each stimulation phase) and after each stimulation phase (high and low intensity; 14 days stimulation each). Stimulation-induced changes in blood parameter will be compared between high and low intensity stimulation.
Stimulation-induced mid-term changes in triglycerides | Baseline (immediately before each stimulation phase), immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  Triglycerides will be assessed at baseline (before each stimulation phase) and after each stimulation phase (high and low intensity; 14 days stimulation each). Stimulation-induced changes in blood levels will be compared between high and low intensity stimulation.
Stimulation-induced mid-term changes in insulin sensitivity | Baseline (immediately before each stimulation phase), immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  Insulin, fasting glucose, and Homeostasis Model Assessment (HOMA-Index) will be assessed at baseline (before each stimulation phase) and after each stimulation phase (high and low intensity; 14 days stimulation each). Stimulation-induced changes in blood parameter will be compared between high and low intensity stimulation.
Stimulation-induced mid-term changes of HbA1c | Baseline (immediately before each stimulation phase), immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  HbA1c will be assessed at baseline (before each stimulation phase) and after each stimulation phase (high and low intensity; 14 days stimulation each). Stimulation-induced changes of HbA1c will be compared between high and low intensity stimulation.
Stimulation-induced mid-term changes in resting heart rate | Baseline (immediately before each stimulation phase), immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  Resting heart rate (HR) will be assessed at baseline (before each stimulation phase) and after each stimulation phase (high and low intensity; 14 days stimulation each). Stimulation-induced changes in HR will be compared between high and low intensity stimulation.
Stimulation-induced mid-term changes in blood pressure | Baseline (immediately before each stimulation phase), immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  Blood pressure (BP) will be assessed at baseline (before each stimulation phase) and after each stimulation phase (high and low intensity; 14 days stimulation each). Stimulation-induced changes in BP will be compared between high and low intensity stimulation.
Stimulation-induced mid-term changes in blood leptin levels | Baseline, immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  The investigators will determine blood leptin levels at baseline and after each stimulation phase (high and low intensity; 14 days stimulation each). Stimulation-induced changes in blood levels will be compared between high and low intensity stimulation.
Stimulation-induced mid-term changes in blood adiponectin levels | Baseline, immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  The investigators will determine blood adiponectin levels at baseline and after each stimulation phase (high and low intensity; 14 days stimulation each). Stimulation-induced changes in blood levels will be compared between high and low intensity stimulation.
Stimulation-induced mid-term changes in blood ghrelin levels | Baseline, immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  The investigators will determine the levels of ghrelin in the blood at baseline and after each stimulation phase (high and low intensity; 14 days stimulation each). Stimulation-induced changes in blood levels will be compared between high and low intensity stimulation.
Stimulation-induced mid-term changes in the levels of Glucagon-like Peptide-1 in the blood | Baseline, immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  The investigators will determine the levels of Glucagon-like Peptide-1 at baseline and after each stimulation phase (high and low intensity; 14 days stimulation each). Stimulation-induced changes in blood levels will be compared between high and low intensity stimulation.
Stimulation-induced mid-term changes in dendrite density as assessed using fiber fraction (anisotropic DBSI-FF) | Baseline, immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  Axonal/dendrite density will be assessed using fiber fraction calculated from DTI images acquired using a 3T Siemens Scanner. Regions of Interest (ROI) will be defined using the Harvard Oxford extended Atlas. Regions of interest include the putamen, caudate, pallidum, and NAcc as well as the hypothalamus. Fiber fraction will be assessed at baseline and after each stimulation phase (high and low intensity; 14 days stimulation each) and compared in predefined ROIs between high and low intensity stimulation.
Stimulation-induced changes in subjective control over eating behaviour | During intervention phase: 14 days
  EMA will be used to assess subjective control over eating behaviour using e.g. the following question: "While you were eating, to what extent did you feel a sense of loss of control?" daily during the intervention phase. Stimulation-induced changes in subjective control over eating behaviour during the intervention phase will be compared between high and low intensity stimulation.
Stimulation-induced mid-term changes in neural response to feedback | Baseline, immediately after the first 14-day stimulation phase and before a 7-day washout, immediately after the second 14-day stimulation phase
  To evaluate neural reward responses, the investigators will assess fMRI bold signals while the earned rewards are displayed during the EAT using a 3T Siemens Scanner. Contrast estimates will include reward magnitude (high, low) and difficulty (high, low) to explore condition specific effects. Region of Interest (ROI) will be defined using the Harvard Oxford extended Atlas. Regions of interest include VTA/SN, caudate, putamen, and NAcc. fMRI metrics will be assessed at baseline and after each stimulation phase (high and low intensity; 14 days stimulation each). Stimulation-induced changes in bold signals will be compared between high and low intensity stimulation.
Stimulation-induced mid-term changes in decision-making between two options of food | During intervention phase: 14 days
  Participants will be asked to rate standardized pictures of food from Charbonnier et al. (2016) in regard to liking, wanting, healthiness, and environmental sustainability at baseline. A choice task will be used to assess changes in decision-making when either two options that have similar values on one dimension (e.g. liking) are presented throughout the intervention phase. Decision weights for the remaining three domains will be estimated and compared between high and low intensity stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Section of Medical Psychology, Department of Psychiatry & Psychotherapy, Faculty of Medicine, University of Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: Yes
After the publication of the key results of the study, all anonymized imaging data will be made publicly available (e.g., at openfmri.org)
Time Frame: Data will become available after an embargo period of 12 months after completion of the study
Access Criteria: Until the data is publicly available, researchers may contact the lead PI to gain access.
URL: http://neuromadlab.com

REFERENCES:
- [Background] Samara A, Li Z, Rutlin J, Raji CA, Sun P, Song SK, Hershey T, Eisenstein SA. Nucleus accumbens microstructure mediates the relationship between obesity and eating behavior in adults. Obesity (Silver Spring). 2021 Aug;29(8):1328-1337. doi: 10.1002/oby.23201. Epub 2021 Jul 5. PMID 34227242
- [Background] Neuser MP, Teckentrup V, Kuhnel A, Hallschmid M, Walter M, Kroemer NB. Vagus nerve stimulation boosts the drive to work for rewards. Nat Commun. 2020 Jul 16;11(1):3555. doi: 10.1038/s41467-020-17344-9. PMID 32678082
- [Background] Charbonnier L, van Meer F, van der Laan LN, Viergever MA, Smeets PAM. Standardized food images: A photographing protocol and image database. Appetite. 2016 Jan 1;96:166-173. doi: 10.1016/j.appet.2015.08.041. Epub 2015 Sep 4. PMID 26344127